CLINICAL TRIAL: NCT07152210
Title: Clinical Study Evaluating the Safety and Preliminary Efficacy of CDH17/GUCY2C CAR-T in the Treatment of Patients With Advanced Colorectal Cancer
Brief Title: Clinical Study on the Safety and Preliminary Efficacy of CDH17/GUCY2C CAR-T in the Treatment of Patients With Advanced Colorectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Bio-gene Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CF-24-008
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer (CRC)
Keywords: Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T (Experimental): The dosage range of 1.0 × 10^6/kg (± 20%) to 5.0 × 10^6/kg (± 20%) of CAR-T cells, administered either intravenously or intratumorally.
  Interventions: Biological: CAR-T

INTERVENTIONS:
Biological: CAR-T — Eligible subjects who successfully passed screening will receive CAR-T cell infusion on Day 0 after lymphodepleting preconditioning chemotherapy.

SUMMARY:
This study is a single-arm, single-center investigator-initiated trial (IIT) designed to evaluate the safety and preliminary efficacy of CDH17/GUCY2C CAR-T cell therapy in patients with advanced colorectal cancer, as well as to assess its pharmacodynamic (PD) and pharmacokinetic (PK) profiles.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this trial, sign the informed consent form.
2. Advanced colorectal cancer patients who have either failed standard treatment, experienced intolerable toxicity, or are unsuitable or unwilling to undergo standard treatment, and voluntarily agree to receive the current treatment.
3. Be able to provide immunohistochemical (IHC) test results from the past 2 years, indicating positive expression of CDH17/GUCY2C targets in tumor tissues.
4. Have at least one extracranial, measurable/assessable lesion according to RECIST 1.1 criteria.
5. Have an ECOG (Eastern Cooperative Oncology Group) performance status score of 0-1 and an expected survival duration of at least 3 months.
6. Have recovered from the toxicity associated with previous treatments, with a CTCAE toxicity grade of less than 2.
7. Have no significant hematopoietic dysfunction and possess adequate organ function.
8. Be able to meet the research center's requirements for apheresis/peripheral blood collection upon successful screening, or have acceptable stored blood cell separation products available.

Exclusion Criteria:

1. Patients who have had or currently have other malignant tumors within the past five years.
2. Presence of brain metastasis.
3. History of clinically significant central nervous system disorders, either in the past or at screening.
4. Imaging indicating tumor invasion of major blood vessels or indistinct borders with blood vessels.
5. Individuals who have received cytotoxic drugs or other interventions, assessed by the investigator as potentially impacting lymphocyte expansion, within 14 days or at least five half-lives (whichever is shorter) prior to blood collection for CAR-T preparation.
6. Presence of other viremias.
7. History of severe allergies.
8. Patients with severe cardiac disease.
9. Patients with severe hepatic and renal dysfunction or disorders of consciousness.
10. Patients with active autoimmune or inflammatory diseases.
11. Patients with objective evidence of past or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-induced pneumonia, severe lung function impairment, etc.
12. Patients who have undergone or are awaiting organ transplantation.
13. Infections requiring intravenous antibiotic therapy for control or are uncontrollable.
14. Individuals who have received live (attenuated) virus vaccines within four weeks prior to screening.
15. Alcoholics or individuals with a history of substance abuse.
16. Pregnant or lactating women.
17. Individuals who have participated in other clinical trials involving drugs within the past 30 days.
18. Patients who, based on the investigator's judgment and/or clinical standards, have contraindications to any study procedures or present other medical conditions that may pose unacceptable risks.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Safety | Up to 1 year after CAR-T infusion
  Count the Incidence of adverse events
Effectiveness evaluation | Up to 1 years after CAR-T infusion
  In accordance with the RECIST 1.1 criteria for assessing the efficacy of solid tumors, the objective response rate (ORR), encompassing patients achieving complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Pharmacokinetic parameters | Up to 1 year after CDH17/GUCY2C CAR-T infusion
  The highest concentration of CAR-T cell expansion in peripheral blood after administration
Pharmacodynamic parameters | Up to 1 year after CAR-T infusion
  The peak values of CAR-T-related cytokines, which include at least IL-6 and IFN-γ.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongguan Taixin Hospital, Dongguan, Guangdong, China

IPD SHARING:
Plan to Share IPD: No